CLINICAL TRIAL: NCT06846190
Title: Effects of Modified Constraint Induced Movement Therapy Versus Virtual Reality Training in Children With Hemiplegic Cerebral Palsy
Brief Title: Modified Constraint Induced Movement Therapy Versus Virtual Reality Training in Children With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR/AHS/22/maria amjad
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: Cerebral palsy; Hemiplegic; Modified constraint induced movement therapy; Spastic; Virtual reality
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: A Randomized clinical trial performed, in which 20 hCP children with the age of 5-16 years will be taken randomly after screening and meeting inclusion criteria. Children will be divided in two groups. Group 1 will receive mCIMT for 5 hours in a day with alternating 3 days a week. Group 2 will receive VR for 25 min in a day with alternating 3 days a week. Pre values were taken at 1st week and then after 4th week mid values of interventions will be taken and post values of intervention will be taken after 8th week of intervention to measure the effects of both therapies.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mCIMT group (Experimental): Clinical experimental: For group -I mCIMT at least 5 waking hours daily for 4 weeks 3 times per week during a 4-week period.
  Interventions: Other: mCIMT
- VR Group (Active Comparator): Clinical experimental: For group -II VR 25 minutes of VR program, every other day, 3 times per week for 4 weeks.
  Interventions: Other: VR

INTERVENTIONS:
Other: mCIMT — mCIMT+ Hot pack will be applied and unaffected hand will be immobilized by a volar resting splint extending from finger tips to the proximal forearm. Use splint every day for at least 5 waking hours daily for 4 weeks and perform daily activities. Program of mCIMT every other day, 3 times per week during a 4-week period.
  Arms: mCIMT group
Other: VR — VR+ Hot pack will be applied. 25 minutes of VR program, every other day, 3 times per week for 4 weeks. Each VR session continued for 10 minutes then 5 minutes rest after that again 10 minutes VR session will do.
  Arms: VR Group

SUMMARY:
Children with hemiplegic cerebral palsy (CP) are characterized by motor impairments mainly lateralized to one side of the body, with greater upper limb than lower limb involvement; these impairments may further limit the daily activities and school participation of children with hemiplegic CP. For the improvement of activity limitations in hemipelagic cerebral palsy children will take 20 hemiplegic cerebral palsy children with the age of 5-16 year all participants will be randomly assign and use modified Constraint induced movement therapy and virtual reality techniques.

mCIMT and Hot pack will be given to group I and unaffected hand will immobilized by a volar resting splint extending from finger tips to the proximal forearm. Use splint every day for at least 5 waking hours individualized, 18-hour program of mCIMT every other day, 3 times per week during a 4-week period. Each modified CIMT session continued for 1.5 hours will give to group I on the other hand VR and Hot pack will give to group II and 18-hour VR program, every other day, 3 times per week for 4 weeks will give Each VR session continued for 1.5 hours. Then evaluate both groups on follow up.

All the data will be collected from Rising Sun Institute by using ABILHAND-KIDS questionnaire and Children's hand-use experience questionnaire. The reliability and validity of tools and mentioned.

The duration of study will be 6-months. Data will be analyzed with the help of SPSS 27

ELIGIBILITY:
Inclusion Criteria:

* Age range between 5 to 16 years of age.
* Medical diagnosis of spastic hemiparetic CP.
* At least 20◦wrist and 10◦ active finger extension from full flexion.
* More movement deficits in 1 upper extremity (less than 2.5 on the Amount of Use scale (AOU) on the Pediatric Motor Activity Log (PMAL)).
* Muscle tone less than 3 on the Modified Ashworth Scale.
* Normal or corrected-to-normal vision and hearing.
* Classified level I, II, or III of the Manual Ability Classification System ( MACS) for Children with CP

Exclusion Criteria:

* Health problems not associated with CP.
* Seizure hemispatial neglect.
* Orthopaedic surgery on the involved upper extremity.
* Botulinum toxin therapy for the affected upper extremity within the past 6 months or within the study period.
* Balance problems

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
CHEQ (Children's hand-use experience questionnaire) | Baseline, 4th week and 8th week
  CHEQ has been developed to capture children's perceived quality of performance when using the affected hand in these situations. CHEQ is an internet-based questionnaire containing 29 items (bimanual activities) presented one by one in random order. Test-retest reliability for the three CHEQ scale was: grasp efficacy, ICC=0.91; time taken, ICC=0.88; and feeling bothered, ICC=0.91. Total Maximum score of each component (quality, duration & psycho-status) was 100 and total maximum score of hand use was 27. Higher the results showed improvement in hand function
ABILHAND-KIDS questionnaire | Baseline, 4th week and 8th week
  ABILHAND-KIDS questionnaire is a valuable tool to assess a child's unimanual and bimanual upper limb activities. The reliability of the ABILHANDS-Kids is good across different observers as a performance- and capacity-based rating method. Test-retest reliability was 0.92. Total Maximum score was 42, mid score was 21 and minimum score was 0. Higher scores showed improvement in activity level of hand use

CONTACTS AND LOCATIONS:
Overall Officials: Maria Amjad, MS-PPT, Principal Investigator — Riphah International University
Locations (1):
- Rising Sun Institute, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roberts H, Shierk A, Clegg NJ, Baldwin D, Smith L, Yeatts P, Delgado MR. Constraint Induced Movement Therapy Camp for Children with Hemiplegic Cerebral Palsy Augmented by Use of an Exoskeleton to Play Games in Virtual Reality. Phys Occup Ther Pediatr. 2021;41(2):150-165. doi: 10.1080/01942638.2020.1812790. Epub 2020 Sep 7. PMID 32892679
- [Background] Wu J, Loprinzi PD, Ren Z. The Rehabilitative Effects of Virtual Reality Games on Balance Performance among Children with Cerebral Palsy: A Meta-Analysis of Randomized Controlled Trials. Int J Environ Res Public Health. 2019 Oct 28;16(21):4161. doi: 10.3390/ijerph16214161. PMID 31661938
- [Background] Aran OT, Sahin S, Kose B, Agce ZB, Kayihan H. Effectiveness of the virtual reality on cognitive function of children with hemiplegic cerebral palsy: a single-blind randomized controlled trial. Int J Rehabil Res. 2020 Mar;43(1):12-19. doi: 10.1097/MRR.0000000000000378. PMID 31658111
- [Background] Simon-Martinez C, Mailleux L, Ortibus E, Fehrenbach A, Sgandurra G, Cioni G, Desloovere K, Wenderoth N, Demaerel P, Sunaert S, Molenaers G, Feys H, Klingels K. Combining constraint-induced movement therapy and action-observation training in children with unilateral cerebral palsy: a randomized controlled trial. BMC Pediatr. 2018 Jul 31;18(1):250. doi: 10.1186/s12887-018-1228-2. PMID 30064396
- [Background] Harb A, Margetis K, Kishner S. Modified Ashworth Scale. 2025 Apr 4. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK554572/ PMID 32119459